CLINICAL TRIAL: NCT05260931
Title: Fetal Cardiac Remodeling in Gestational Diabetic Pregnancies at the Moment of Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med Flavio Hernández Castro, Dr. med Flavio Hernández Castro, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: GI18-0012
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Fetal Cardiac Anomaly; Gestational Diabetes
Keywords: Fetal heart; Cardiac remodeling; Gestational diabetes; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes group: This group will be formed by women with gestational diabetes (GD). The diagnosis of GD was made when one or more of the venous plasma glucose measurements met or exceeded the following thresholds after a 75 g Oral Glucose Tolerance Test (75 g OGTT): fasting blood glucose ≥ 92 mg/dL, 1 h plasma glucose level ≥ 180 mg/dL or 2 h plasma glucose level ≥ 153 mg/dL, as recommended by the International Association of the Diabetes and Pregnancy Study Groups.
  Interventions: Diagnostic Test: Fetal echocardiography
- Control group: This group will be formed by women with normal 75 g OGTT findings.
  Interventions: Diagnostic Test: Fetal echocardiography

INTERVENTIONS:
Diagnostic Test: Fetal echocardiography — Two-dimensional, M mode, and Doppler echocardiographic examination performed to rule out cardiac defects and to evaluate cardiac morphometry and function. Cardiac, thoracic, and ventricular areas and diameters measured on 2-dimensional images from an apical or basal four-chamber (4 ChV) view at end diastole. Ventricular sphericity indices calculated by dividing the longitudinal by basal-transverse ventricular diameters. Atrial areas at maximum distension at end of systole. Atria and ventricle to-heart ratios calculated. Myocardial wall thicknesses and ventricular shortening/ejection fractions obtained from M-mode transverse 4 ChV. MAPSE/TAPSE assessed by M-mode from an apical or basal 4 ChV. Mitral and tricuspid early and late ventricular filling obtained by Doppler, and E/A ratios calculated. Left and right myocardial performance indices obtained from Doppler spectrum in a cross-sectional image of the thorax.

SUMMARY:
The aim of the present study will be to evaluate whether fetal cardiac remodeling is already present at the moment of the diagnosis of gestational diabetes (GD) in comparison with fetuses of healthy pregnant women.

DETAILED DESCRIPTION:
We will recruited patients at the time of 75-g oral glucose tolerance test (OGTT); GDM will be diagnosed at 24-28.6 weeks when one or more of the venous plasma glucose measurements met or exceeded the following thresholds: fasting blood glucose ≥ 92 mg/dL; 1 h plasma glucose level ≥ 180 mg/dL; or 2 h plasma glucose level ≥ 153 mg/dL, as recommended by the International Association of the Diabetes and Pregnancy Study Groups. Consecutive women with singleton pregnancies with negative OGTT findings wil be also recruited during this period.

Maternal Characteristics The baseline variables, including maternal age, height, weight (1st ans 2nd trimester), parity will be collected at the time of the ultrasound examination. Additionally, fasting blood glucose, 1 h plasma glucose level and 2 h plasma glucose level in 75-g OGTT and glycated hemoglobin A1 (HbA1c) will be recorded. Body mass index of all mothers will be calculated.

Ultrasonographic examination using Voluson E6 (GE Medical Systems, Milwaukee, MI, USA) with 2-8 MHz linear curved-array probes, including estimated fetal weight, anomaly scan, and fetal echocardiography. The images will be recorded as clips and anonymized, and all the measurements will be performed offline.

Fetal biometric measurements will be obtained following ISUOG recommendations and fetal weight with Hadlock 4 formula.

Comprehensive two-dimensional, M-mode, and Doppler echocardiographic examination will be performed to rule out cardiac defects, and to evaluate cardiac morphometry and function following standard protocols. Cardiac, thoracic, and ventricular areas and diameters will be measured on 2-dimensional images from an apical or basal four-chamber (4 ChV) view at end diastole. Ventricular sphericity indices calculated by dividing the longitudinal by basal-transverse ventricular diameters. Atrial areas measured at maximum distension at end of systole. Atria and ventricle to-heart ratios will be calculated. Myocardial wall thicknesses measured on M-mode images from a transverse 4 ChV. Ventricular ejection fractions will be obtained from M-mode transverse 4 ChV using the Teichholz's formula. MAPSE/TAPSE will be assessed by M-mode from an apical or basal 4 ChV. Mitral and tricuspid early and late ventricular filling will be obtained by Doppler, and E/A ratios calculated. The left and right myocardial performance indices obtained from Doppler spectrum in a cross-sectional image of the thorax.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who will undergo 75g OGTT between 24 and 28.6 weeks of gestation will be invited to participate. Before being recruited, the objective of the research will be explained, the confidential nature of the information and informed consent will be requested. Inclusion criteria: singleton spontaneously conceived pregnancy, first trimester ultrasound screening to establish gestational age and first trimester serum glycemia < 92 mg/dL.

Exclusion Criteria:

* Those women with conditions or comorbidities that could induce cardiac remodeling and suboptimal function or could modify fetal growth will be excluded: fetus conceived by ssisted reproductive technology, pregestational diabetes, systemic lupus erythematosus, antiphospholipid antibody syndrome and other thrombophilias, heart disease, chronic pulmonary or renal disease, and thyroid disease. In addition, any hypertensive disease in pregnancy or derived complications (chronic arterial hypertension, gestational hypertension, pre-eclampsia, eclampsia). Patients with exposure to substances that could affect fetal weight will be excluded: teratogens (cyclophosphamide, valproic acid, antithrombotic drugs), tobacco, alcohol, cocaine or coffee consumption of more than 1 cup/day. Finally, women with a history of intrauterine growth restriction (IUGR) and/or preeclampsia in previous pregnancies, high risk of IUGR and/or preeclampsia in the current pregnancy estimated at first trimester screening, mean uterine artery greater than the 95th percentile for gestational age at 24-28.6 weeks, fetal structural defects or markers of aneuploidy on first or second trimester ultrasonography will be also excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: The study population will consist of patients with singleton spontaneously conceived pregnancies who will undergo 75g OGTT at 24-28.6 weeks, with regular medical checkups throughout their entire pregnancy, delivered after 24-week gestation and fulfilled inclusion criteria. This study will be performed according to the standards of the Helsinki Declaration and approval will be obtained from the ethics and educational issues coordinating committee of our University Hospital.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-05 (Estimated)

PRIMARY OUTCOMES:
Ventricular sphericity indices | 45-60 minutes
  Left and right Ventricular sphericity indices will be calculated by dividing the longitudinal by basal-transverse ventricular diameters on 2-dimensional images from an apical or basal four-chamber (4 ChV) view at end diastole.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Hernández Castro, MD PhD, Principal Investigator — Hospital Universitario UANL
Locations (1):
- Hospital Universitario "Dr. José E. González" UANL, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No